CLINICAL TRIAL: NCT02926001
Title: Empirical Evaluation of the Short Term Impact of a Sugar-Sweetened Beverage Tax in Chile
Brief Title: Evaluation of the Impact of a Sugar-Sweetened Beverage Tax in Chile
Status: Completed | Type: Observational
Sponsor: Marc Suhrcke (Other)
Collaborators: University of Chile (Other)
Responsible Party: Sponsor-Investigator, Marc Suhrcke, Professor, University of York
Organization: University of York (Other)
Other Study IDs: MR/N026640/1
Record Dates: First submitted 2016-10-04; First posted 2016-10-06 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Disease; Obesity
Keywords: Taxes; Beverages/economics; Carbonated Beverages/economics; Diet, Food and Nutrition/economics; Economics; Energy Intake; Risk Factors
MeSH Terms: conditions — Chronic Disease; Obesity

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate formally the short term impacts of the tax policy applied to Sugar-Sweetened Beverages (SSBs) in Chile. The Impuesto Adicional a las Bebidas Analcohólicas (IABA, or "additional tax on soft drinks") in Chile was enacted in October 2014, affecting any non-alcoholic beverages to which colorants, flavourings or sweeteners have been added. For beverages above an added sugar concentration of at least 6.25 grams per 100ml (or equivalent proportion), the tax was increased from 13% to 18%, while for those below this threshold the tax was decreased to 10%, producing an 8% tax difference between these beverage groups. This impact evaluation analysis of the Chilean sugar-sweetened beverage (SSB) tax will estimate the impact of increasing the tax as well as decreasing the tax on soft drinks. The study will use household level grocery purchasing data for Chile. The purchasing records are available from October 2011 to September 2015 (three years before; and one year after the implementation of the tax in October 2014). The investigators will use a series of quasi-experimental approaches to evaluate the causal impact of the SSB tax policy on consumers' behaviour as well as on industry responses in the form of pricing and price promotion decisions.

ELIGIBILITY:
Inclusion Criteria:

* Household in Chile that agreed to participate in the purchasing survey and provided data to a satisfactory degree for the first 2 months.

Exclusion Criteria:

* Households that are unwilling to participate in the survey. Households that change physical address. Households with poor compliance to the survey.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population is 2,836 households that arenationally representative of urban areas in Chile.
Sampling Method: Probability Sample
Enrollment: 2836 (Actual)
Dates: Start 2011-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Volume of sugar-sweetened beverage purchased | October 2011 - September 2015

SECONDARY OUTCOMES:
Consumer shopping patterns - Frequency | October 2011 - September 2015
  Frequency of Purchasing
Consumer shopping patterns - Volume | October 2011 - September 2015
  Volume of Purchases
Market price of sugar-sweetened beverages | October 2011 - September 2015
Body mass index of household members | October 2011 - September 2015

CONTACTS AND LOCATIONS:
Overall Officials: Marc Suhrcke, PhD, Principal Investigator — Centre for Health Economics, University of York; Ryota Nakamura, PhD, Principal Investigator — Centre for Health Economics, University of York; Andrew J Mirelman, PhD, Principal Investigator — Centre for Health Economics, University of York; Cristobal Cuadrado, MD, PhD, Principal Investigator — University of Chile; Nicolas Silva, MD, Principal Investigator — University of Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nakamura R, Mirelman AJ, Cuadrado C, Silva-Illanes N, Dunstan J, Suhrcke M. Evaluating the 2014 sugar-sweetened beverage tax in Chile: An observational study in urban areas. PLoS Med. 2018 Jul 3;15(7):e1002596. doi: 10.1371/journal.pmed.1002596. eCollection 2018 Jul. PMID 29969456